CLINICAL TRIAL: NCT00645385
Title: Treatment Of Newly Diagnosed, High-Grade, Malignant Glioma With Polifeprosan 20 Containing Carmustine Implant (Gliadel® Wafer) Using MR Spectroscopy Data As A Primary Indicator Of Therapeutic Response.
Brief Title: Examination of Changes on Magnetic Resonance Imaging (MRI) and Magnetic Resonance Spectroscopy (MRS) in Patients Who Receive Gliadel Wafers During Initial Surgery for Glioblastoma Multiforme. Response or Failure to Gliadel Wafers for Subjects With Glioblastoma Multiforme.
Acronym: Gliadel-MRS
Status: Withdrawn | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 07090991
Record Dates: First submitted 2008-03-20; First posted 2008-03-27 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma
Keywords: GBM; AA; AO; Brain; Tumors; Malignant; Glioblastoma; Multiforme; Carmustine; implant; BCNU; Gliadel; Wafers; MRS; Spectroscopy
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Neoplasms | interventions — Proton Magnetic Resonance Spectroscopy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRS of the neural system: MRS to study epilepsy, Alzheimer's disease, brain tumors, and the effects of drugs on brain growth and metabolism.
  Interventions: Other: MRS Spectroscopy

INTERVENTIONS:
Other: MRS Spectroscopy — Magnetic Resonance Spectroscopy uses a continuous band of radio wave frequencies to excite hydrogen atoms in a variety of chemical compounds other than water. These compounds absorb and emit radio energy at characteristic frequencies, or spectra, that can be used to identify them. Generally, a color image is created by assigning a hue to each distinctive spectral emission. This comprises the "spectroscopy" part of MRS. MRS is still experimental, and is available in only a few research centers.
  Physicians mainly use MRS to study the brain and disorders such as epilepsy, Alzheimer's disease, brain tumors, and the effects of drugs on brain growth and metabolism. The technique is also useful in evaluating metabolic disorders of the muscles and nervous system. MRS is a noninvasive scan similar to an MRI that may be done at the same time as an MRI.
  Other Names: MRS; Magnetic Resonance Spectroscopy

SUMMARY:
Subjects with newly diagnosed brain tumors who undergo surgical resection and whose pathology in the operating room shows a high grade glioma will be eligible.

During a screening visit, the study will be discussed, inform consent discussed and signed, a medical history will be taken and a physical examination and laboratory tests will be performed. If these tests are all within acceptable ranges, the subject will be considered for inclusion on this treatment protocol. If the results of any tests are extremely different from normal expected values, she/he may not be able to participate.

Prior to surgery, the subject will have a contrast enhanced MRI and MRS. The neurosurgeon will attempt to remove the majority of the tumor in the operating room and will send a portion of the specimen removed to the pathologist immediately. This is called a "frozen section". If the pathologist believes that the tumor is a high-grade malignant brain tumor, then the surgeon will place up to 8 dime-sized chemotherapy wafers in the tumor cavity of the brain. The remainder of the tumor specimen will be given to the pathologist to review more closely in the laboratory. If the frozen section does not show that the tumor is a high-grade malignant brain tumor, the subject will not receive the Gliadel wafers and will be removed from the study. The surgeon will then discuss with the subject the appropriate treatment options for the disease he or she has.

During recovery in the hospital, another contrast enhanced MRI will be performed within the first 72 hours after surgery. This is a standard of care for patients who are not involved on this protocol as well. The subject will have another contrast enhanced MRI and MRS performed at the 21st Day after his or her surgery. After Day 21, He or she may begin other forms of treatment. The last contrast enhanced MRI and MRS assessment will be performed 12 weeks after the surgery and the implantation of the Gliadel wafers. Further MRI and MRS may be performed subsequently at the discretion of the doctor.

Throughout the course of treatment, clinical data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of >17 years of age.
* Patients with a documented histologic diagnosis of high grade malignant glioma on intraoperative frozen section or squash preparation.
* Solitary, supratentorial lesions that do not cross the midline
* Patients must have a Karnofsky performance status >=60% (or the equivalent ECOG level of 0-2) (see Appendix A; Performance Status Evaluation) and an expected survival of > three months.
* Patients must have adequate hematologic reserve with WBC>=3000/mm3, absolute neutrophils >=1500/mm3 and platelets >=100,000/ mm3.
* Pre-enrollment chemistry parameters must show: bilirubin<1.5X the institutional upper limit of normal (IUNL); AST or ALT<2.5X IUNL and creatinine<1.5X IUNL.
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study.
* Patients must be able to understand and give written informed consent. Informed consent must be obtained at the time of patient screening.

Exclusion Criteria:

* Known hypersensitivity or allergy to BCNU (carmustine) or other components of the Gliadel® wafer, such as polifeprosan polymer.
* Multifocal CNS disease
* Diagnosis of prior CNS tumor
* Women who are pregnant or lactating.
* Posterior Fossa or Brain stem tumor
* Open communication of the resection cavity with the ventricular system and tumors that cross the midline.
* Concurrent severe medical (e.g., active infection, acute hepatitis, cardiac arrhythmia, unstable angina, congestive heart failure, uncontrolled diabetes mellitus, uncontrolled seizures, pulmonary insufficiency, pulmonary fibrosis, pulmonary embolus, etc) or psychiatric illness, or abnormal laboratory values that preclude surgical candidacy or limits expected survival to less than 12 weeks. If in doubt, contact the Study Principal Investigator.
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06-01 (Actual); Study Completion 2011-06-01 (Actual)

PRIMARY OUTCOMES:
Stabilization or reduction of tumor on gadolinium enhanced MRI and changes in choline/creatine ratio and NAA on MR Spectroscopy | June 2011

SECONDARY OUTCOMES:
Median survival, 6-month survival, and progression free survival. | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Susan C. Pannullo, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College Department of Neurosurgery, New York, New York, United States